CLINICAL TRIAL: NCT02384850
Title: An Investigator Initiated Phase 1 Trial To Evaluate mFOLFOX6 With Selinexor (KPT-330), An Oral Selective Inhibitor Of Nuclear Export (SINE), In Patients With Metastatic Colorectal Cancer
Brief Title: Phase 1 Trial To Evaluate mFOLFOX6 With Selinexor In Patients With Metastatic Colorectal Cancer
Acronym: SENTINEL
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: GSO Global Clinical Research BV (Other)
Collaborators: Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SENTINEL
Record Dates: First submitted 2015-03-02; First posted 2015-03-10 (Estimated); Results first posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-02

CONDITIONS: Colorectal Neoplasm
Keywords: metastatic
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — selinexor; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Intervention Model Description: Dose level 1: Oxaliplatin at a dose of 85 mg/m2 IV over two hours (Day 1) 5-FU 400 mg/m2 IV bolus (Day 1) Leucovorin 400 mg/m2 IV over two hours (Day 1) 5-FU 2400 mg/m2 IV over 46 hours (Day 1-3) Selinexor 40 mg, PO (Day 1, 3 and 8) Dose level 2: Oxaliplatin at a dose of 85 mg/m2 IV over two hours (Day 1) 5-FU 400 mg/m2 IV bolus (Day 1) Leucovorin 400 mg/m2 IV over two hours (Day 1) 5-FU 2400 mg/m2 iv over 46 hours (Day 1-3) Selinexor 60 mg, PO (Day 1, 3 and 8) Dose level 3: Oxaliplatin at a dose of 85 mg/m2 iv over two hours (Day 1) 5-FU 400 mg/m2 iv bolus (Day 1) Leucovorin 400 mg/m2 iv over two hours (Day 1) 5-FU 2400 mg/m2 iv over 46 hours (Day 1-3) Selinexor 80 mg, PO (Day 1, 3 and 8) Dose level -1: Oxaliplatin at a dose of 85 mg/m2 IV over two hours (Day 1) 5-FU 400 mg/m2 IV bolus (Day 1) Leucovorin 400 mg/m2 IV over two hours (Day 1) 5-FU 2400 mg/m2 IV over 46 hours (Day 1-3) Selinexor 20 mg, PO (Day 1, 3 and 8)
Oversight: Data Monitoring Committee: No

ARMS (1):
- Selinexor + mFOLFOX6 (Experimental): Different Dose Levels of Selinexor will be evaluated in combination with mFOLFOX6 (see interventions)
  Interventions: Drug: Selinexor; Drug: Oxaliplatin; Drug: 5-FU; Drug: Folinic Acid

INTERVENTIONS:
Drug: Selinexor — Dose Level 1: 40 mg on day 1, 3 and 8 in a two-weeks cycle. Dose Level 2: 60 mg on day 1, 3 and 8 in a two-weeks cycle. Dose Level 3: 80 mg on day 1, 3 and 8 in a two-weeks cycle. Dose Level -1: 20 mg on day 1, 3 and 8 in a two-weeks cycle.
  Other Names: KPT-330
Drug: Oxaliplatin — 85 mg/m² IV over 2 hours, Day 1 of a two-weeks cycle
  Other Names: oxalatoplatin
Drug: 5-FU — 400 mg/m² IV bolus, Day 1 of a two-weeks cycle 2,400 mg/m² continuous infusion IV, Days 1-3
  Other Names: 5-fluorouracil
Drug: Folinic Acid — 400 mg/m2 IV over 2 hours, Day 1 of a two-weeks cycle
  Other Names: leucovorin

SUMMARY:
This trial will evaluate the combination treatment of established chemotherapy regimen mFOLFOX6 with Selinexor, an oral Selective Inhibitor Of Nuclear Export, in patients with metastatic Colorectal Cancer. The purpose is to determine the maximum tolerated dose (MTD) of selinexor in combination with mFOLFOX6.

DETAILED DESCRIPTION:
This was a multi center, open-label, non-randomized phase I trial study to determine the MTD of a combination of mFOLFOX6 (Folinic Acid (Leucovorin)-Fluorouracil-Oxaliplatin) and selinexor in patients with metastatic colorectal cancer.

After screening and registration in the study, all enrolled patients were to be treated with oxaliplatin (85 mg/m² IV over 2 hours, Day 1), 5-FU (5-Fluorouracil 400 mg/m2 IV bolus, Day 1), leukovorin (400 mg/m2 IV over 2 hours, Day 1), and 5-FU (2,400 mg/m² continuous infusion, Days 1-3) every 2 weeks and escalating doses of selinexor as follows:

Patients in Dose Level 1 were to receive oral selinexor 40 mg on day 1, 3, and 8.

Patients in Dose Level 2 were to receive oral selinexor 60 mg on day 1, 3, and 8.

Patients in Dose Level 3 were to receive oral selinexor 80 mg on day 1, 3, and 8.

Patients in Dose Level -1 were to receive oral selinexor 20 mg on day 1, 3, and 8.

The MTD was defined as the highest dose level at which six patients had been treated with no toxicity and tolerance of the dose escalation of Selinexor with mFOLFOX6 was evaluated.

Six patients were to be initially treated in a cohort. Safety data were monitored in real time. As soon as last patient of the cohort (either 6th or 9th) reached day 28, safety data of all patients within that cohort were reviewed for decision about opening up a new cohort by moving to the next dose level or expand the cohort or discontinue dose escalation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed diagnosis of colorectal cancer presenting with unresectable stage IV (UICC) disease (primary tumor may be present)
2. Patients who are feasible for treatment with FOLFOX (prior adjuvant or palliative treatment is allowed)
3. ECOG (Eastern Cooperative Oncology Group) Performance status ≤ 1
4. Life expectancy > 3 months
5. Age ≥18 years
6. Haematologic function as follows (5% deviation allowed):

   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * platelets ≥ 100 x109/L
   * hemoglobin ≥ 9 g/dl or 5.59 mmol/l
7. Adequate liver function as follows (10% deviation allowed)

   * serum alanine transaminase (ALT) ≤ 2.5 x ULN (in case of liver metastases < 5 x ULN)
   * total bilirubin ≤ 1.5 x ULN (patients with Gilbert's syndrome total bilirubin ≤2.5 x ULN)
8. Adequate renal function as follows (10% deviation allowed)

   · creatinine ≤ 1.5 x ULN
9. Signed written informed consent
10. Women of child-bearing potential must have a negative pregnancy test

Exclusion Criteria:

adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy; 2. Treatment with any systemic anticancer therapy ≤ 3 weeks prior to cycle 1 day 1 3. Uncontrolled active infection (Hepatitis B and C infection are NOT exclusion criteria) and/or known HIV infection; 4. Renal failure requiring haemodialysis or peritoneal dialysis; 5. Patients who are pregnant or breast-feeding; 6. Patients with significantly diseased or obstructed gastrointestinal tract, malabsorption, uncontrolled vomiting or diarrhea resulting in inability to swallow oral medications; 7. Presence of symptomatic Central nervous system (CNS) metastasis 8. Unresolved toxicity from previous anti-cancer therapy or incomplete recovery from surgery, in particular oxaliplatin-induced peripheral neuropathy > grade 1.

9. Any of the following within the 12 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis, or other thromboembolic event.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-03; Primary Completion 2017-03-09 (Actual); Study Completion 2017-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Bokemeyer, Prof. Dr., Principal Investigator — University Hospital Hamburg
Locations (2):
- University Hospital Antwerpen, Antwerp, Belgium
- University Hospital Hamburg, Hamburg, Germany

REFERENCES:
- [Derived] Nilsson S, Stein A, Rolfo C, Kranich AL, Mann J, Papadimitriou K, Theile S, Amberg S, Bokemeyer C. Selinexor (KPT-330), an Oral Selective Inhibitor of Nuclear Export (SINE) Compound, in Combination with FOLFOX in Patients with Metastatic Colorectal Cancer (mCRC) - Final Results of the Phase I Trial SENTINEL. Curr Cancer Drug Targets. 2020;20(10):811-817. doi: 10.2174/1568009620666200628105727. PMID 32598257

RESULTS

PARTICIPANT FLOW:
Groups:
- Selinexor 40 mg+ mFOLFOX6: Selinexor: Dose Level 1: 40 mg on day 1, 3 and 8 in a two-weeks cycle.
  Oxaliplatin: 85 mg/m² IV over 2 hours, Day 1 of a two-weeks cycle
  5-FU: 400 mg/m² IV bolus, Day 1 of a two-weeks cycle 2,400 mg/m² continuous infusion IV, Days 1-3
  Folinic Acid: 400 mg/m2 IV over 2 hours, Day 1 of a two-weeks cycle
- Selinexor 20mg + mFOLFOX6: Selinexor: Dose Level -1: 20 mg on day 1, 3 and 8 in a two-weeks cycle.
  Oxaliplatin: 85 mg/m² IV over 2 hours, Day 1 of a two-weeks cycle
  5-FU: 400 mg/m² IV bolus, Day 1 of a two-weeks cycle 2,400 mg/m² continuous infusion IV, Days 1-3
  Folinic Acid: 400 mg/m2 IV over 2 hours, Day 1 of a two-weeks cycle
Period: Overall Study
Arm/Group | Selinexor 40 mg+ mFOLFOX6 | Selinexor 20mg + mFOLFOX6
Started | 4 | 6
Completed | 2 | 4
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Selinexor 40mg + mFOLFOX6: Selinexor: Dose Level 1: 40 mg on day 1, 3 and 8 in a two-weeks cycle.
  Oxaliplatin: 85 mg/m² IV over 2 hours, Day 1 of a two-weeks cycle
  5-FU: 400 mg/m² IV bolus, Day 1 of a two-weeks cycle 2,400 mg/m² continuous infusion IV, Days 1-3
  Folinic Acid: 400 mg/m2 IV over 2 hours, Day 1 of a two-weeks cycle
- Total: Total of all reporting groups
Arm/Group | Selinexor 40mg + mFOLFOX6 | Selinexor 20mg + mFOLFOX6 | Total
Number analyzed (Participants) | 4 | 6 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 7
  >=65 years | 0 | 3 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 6 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 0 | 2 | 2
  Germany | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Numbers of Patients With Dose Limiting Toxicities
Description: Primary objective is the determination of the maximum tolerated dose (MTD) of selinexor in combination with mFOLFOX6 in patients with metastatic colorectal cancer.
  Criteria to assess MTD was the experience of AEs > grade 3, discontinuation from study treatment due to adverse events or withdrawal of consent by the patients.
Time Frame: 28 days of treatment
Population: The study was closed due to toxicity despite dose reduction to 20 mg Seiinexor.
Measure: Count of Participants; unit: Participants
Arm/Group | Selinexor 40 mg+ mFOLFOX6 | Selinexor 20mg + mFOLFOX6
Number analyzed (Participants) | 4 | 6
Participants
  Discontinuation due to Adverse events | 2 | 2
  Discontinuation due to Withdrawal of Consent | 2 | 2
  Discontinuation due to Progressive Disease | 0 | 2

2. Secondary Outcome: Overall Response Rate
Description: Secondary objectives are to determine the efficacy and tolerability of selinexor in combination with mFOLFOX6 in patients with metastatic colorectal cancer by
  - Overall response rate (RR) (acc. to RECIST v1.1)
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed byCT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 2 years
Population: Due to the low number of patients, no conclusions can be drawn from analysis of the efficacy data.
Measure: Count of Participants; unit: Participants
Arm/Group | Selinexor 40 mg+ mFOLFOX6 | Selinexor 20mg + mFOLFOX6
Number analyzed (Participants) | 4 | 6
Participants | 0 | 1

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Secondary objectives are to determine the efficacy and tolerability of selinexor in combination with mFOLFOX6 in patients with metastatic colorectal cancer by
  - Progression free survival (PFS) The disease status was measured by CT/MRI and evaluated according to RECIST 1.1 criteria every 8 weeks during treatment, at End of Treatment and every 3 weeks during Follow-up to determine time until patient has Progressive Disease (PD). PD is defined according to RECIST v1.1 at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: 2 years
Population: Four patients withdrew consent to further participate in the study before the first tumour assessment had been performed. No data on PD were available for those patients. Additionally, for two patients in cohort 2, no information on PD during the follow-up period is available.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Selinexor 40 mg+ mFOLFOX6 | Selinexor 20mg + mFOLFOX6
Number analyzed (Participants) | 2 | 2
months | NA (NA) — Based on limited number of participants, the Kaplan-Meier analyses could not be performed as planned. | NA (NA) — Based on limited number of participants, the Kaplan-Meier analyses could not be performed as planned.

4. Secondary Outcome: Number of Patients Still Alive at End of Study (Overall Survival)
Description: Secondary objectives are to determine the efficacy and tolerability of selinexor in combination with mFOLFOX6 in patients with metastatic colorectal cancer by
  - Overall survival (OS)
  Overall survial is defined as length of time from start of treatment that patients are still alive. For this time-to-event variables the Kaplan-Meier method was intended to be used
Time Frame: 2 years
Population: Due to sparse data set, no analysis with Kaplan-Meier methods was done.
Measure: Count of Participants; unit: Participants
Arm/Group | Selinexor 40 mg+ mFOLFOX6 | Selinexor 20mg + mFOLFOX6
Number analyzed (Participants) | 2 | 4
Participants | 0 | 2

5. Secondary Outcome: Number of Patients Experiencing Adverse Events
Description: Secondary objectives are to determine the efficacy and tolerability of selinexor in combination with mFOLFOX6 in patients with metastatic colorectal cancer by
  - Toxicity (acc. to NCI Common Terminology Criteria for Adverse Events (CTC AE) v4.03)
Time Frame: treatment start to up to 30 days after last dose
Population: All 10 patients were treated with at least one dose of Selinexor.
Measure: Count of Participants; unit: Participants
Arm/Group | Selinexor 40 mg+ mFOLFOX6 | Selinexor 20mg + mFOLFOX6
Number analyzed (Participants) | 4 | 6
Participants
  Patients with AEs of any CTCAE Grade | 4 | 6
  Patients with AEs of at least CTCAE Grade 3 | 4 | 6
  Patients with Selinexor related AEs of any Grade | 4 | 4
  Patients with Selinexor related AEs of at least Grade 3 | 4 | 5
  Patients with chemotherapy related AEs of any Grade | 4 | 6
  Patients with chemotherapy related AEs of at least Grade 3 | 4 | 3
  Patients with AEs leading to discontinuation | 2 | 2
  Patients with at least 1 SAE | 2 | 3
  Patients with at least 1 SAE related to Selinexor | 1 | 1
  Patients with at least 1 SAE related to chemotherapy | 1 | 3

ADVERSE EVENTS:
Time Frame: Adverse Events were monitored from the date of informed consent until 30 days after the last dose of study medication (end of treatment visit). Patients who discontinued for reasons other than withdrawal of consent were followed for a maximum of 24 months for progression-free survival and overall survival, so deaths were monitored for up to 2 years for patients in follow-up.
Arm/Group | Selinexor 40mg + mFOLFOX6 | Selinexor 20mg + mFOLFOX6
All-Cause Mortality (participants affected / at risk) | 0/4 | 2/6
Serious Adverse Events (participants affected / at risk) | 2/4 | 3/6
Other Adverse Events (participants affected / at risk) | 4/4 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selinexor 40mg + mFOLFOX6 (N=4) | Selinexor 20mg + mFOLFOX6 (N=6)
PULMONARY EMBOLISM (Vascular disorders) | 1 (1) | 0 (0)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 1 (1)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 (0) | 1 (1)
GENERAL MALAISE (General disorders) | 0 (0) | 1 (1)
SEIZURE (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Selinexor 40mg + mFOLFOX6 (N=4) | Selinexor 20mg + mFOLFOX6 (N=6)
NAUSEA (Gastrointestinal disorders) | 4 (10) | 4 (4)
VOMITING (Gastrointestinal disorders) | 3 (4) | 3 (4)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0)
DIARRHEA (Gastrointestinal disorders) | 3 (4) | 4 (4)
ANEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 5 (5)
HYPONATREMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 1 (1) | 1 (1)
WEIGHT LOSS (Investigations) | 1 (2) | 1 (1)
ANOREXIA (Metabolism and nutrition disorders) | 1 (2) | 3 (3)
ASTHENIA (General disorders) | 1 (3) | 0 (0)
INFECTION OF UNKNOWN ORIGIN (Infections and infestations) | 0 (0) | 1 (3)
DIZZINESS (Nervous system disorders) | 0 (0) | 2 (2)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (1)
INSOMNIA (Psychiatric disorders) | 0 (0) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (2) | 2
BODY PAIN (General disorders) | 0 (0) | 1 (1)
DOUBLE VISION (Eye disorders) | 0 (0) | 1 (1)
PAIN INGUINAL RIGHT (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SENSORY NEUROPATHY (Nervous system disorders) | 0 (0) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 1 (1)
BLURRED VISION (Eye disorders) | 2 (2) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 1 (1)
HEARING IMPAIRMENT (Ear and labyrinth disorders) | 0 (0) | 1 (1)
FLU-LIKE SYMPTOMS (General disorders) | 0 (0) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
MALAISE (General disorders) | 0 (0) | 1 (1)
HYPOKALEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
POLYNEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-01-22): https://cdn.clinicaltrials.gov/large-docs/50/NCT02384850/Prot_SAP_000.pdf